CLINICAL TRIAL: NCT00964951
Title: A Phase II Study in Healthy Adult and Elderly Populations to Assess the Safety and Immunogenicity of a CSL H1N1 Influenza Vaccine Administered at Different Dose Levels Given With and Without GlaxoSmithKline AS03 Adjuvant
Brief Title: CSL H1N1 Influenza Vaccine Administered at Different Dose Levels With and Without AS03 Adjuvant in Healthy Adult and Elderly Populations
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0060; N01AI80007C
Record Dates: First submitted 2009-08-20; First posted 2009-08-25 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2009-10

CONDITIONS: Influenza
Keywords: H1N1, influenza A viruses, vaccine, elderly
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- Group 3: 15 mcg H1N1 vaccine + AS03 adjuvant (Experimental): 150 subjects (100 aged 18-64 and 50 aged greater than or equal to 65) to receive 15 mcg H1N1 vaccine plus AS03 adjuvant on Day 0 and Day 21.
  Interventions: Biological: AS03; Biological: Inactivated H1N1 Vaccine
- Group 1: 3.75 mcg H1N1 vaccine + AS03 adjuvant (Experimental): 150 subjects (100 aged 18-64 and 50 aged greater than or equal to 65) to receive 3.75 mcg H1N1 vaccine plus AS03 adjuvant on Day 0 and Day 21.
  Interventions: Biological: AS03; Biological: Inactivated H1N1 Vaccine
- Group 4: 7.5 mcg H1N1 vaccine unadjuvanted (Experimental): 150 subjects (100 aged 18-64 and 50 aged greater than or equal to 65) to receive 7.5 mcg H1N1 vaccine unadjuvanted on Day 0 and Day 21.
  Interventions: Biological: Inactivated H1N1 Vaccine
- Group 2: 7.5 mcg H1N1 vaccine + AS03 adjuvant (Experimental): 150 subjects (100 aged 18-64 and 50 aged greater than or equal to 65) to receive 7.5 mcg H1N1 vaccine plus AS03 adjuvant on Day 0 and Day 21.
  Interventions: Biological: AS03; Biological: Inactivated H1N1 Vaccine
- Group 5: 15 mcg H1N1 vaccine unadjuvanted (Experimental): 150 subjects (100 aged 18-64 and 50 aged greater than or equal to 65) to receive 15 mcg H1N1 vaccine unadjuvanted on Day 0 and Day 21.
  Interventions: Biological: Inactivated H1N1 Vaccine

INTERVENTIONS:
Biological: AS03 — AS03 adjuvant administered with 3.75, 7.5, or 15 mcg Inactivated H1N1 Vaccine.
  Arms: Group 1: 3.75 mcg H1N1 vaccine + AS03 adjuvant; Group 2: 7.5 mcg H1N1 vaccine + AS03 adjuvant; Group 3: 15 mcg H1N1 vaccine + AS03 adjuvant
Biological: Inactivated H1N1 Vaccine — Inactivated influenza H1N1 vaccine with AS03 adjuvant, delivered intramuscularly (IM) as 3.75, 7.5, or 15 micrograms per dose; and inactivated influenza H1N1 vaccine without adjuvant, delivered intramuscularly as 7.5 or 15 micrograms per dose. All doses of vaccine with or without adjuvant will be administered as a single 0.5 mL IM injection in the deltoid muscle of the preferred arm.

SUMMARY:
The purpose of this study is to see how the body reacts to different strengths of the H1N1 flu shot when it is given with or without an "adjuvant." An adjuvant is a substance that may cause the body to produce more antibodies when it is given with a vaccine. This study will also compare how age affects the body's response to the H1N1 flu shot. In this study, 3 strengths of the H1N1 flu shot will be tested combined with an adjuvant. In addition, 2 strengths of the H1N1 flu shot will be tested without adjuvant. Two H1N1 flu shots of the same strength, with or without adjuvant, will be given about 3 weeks apart. Participants will include up to 800 healthy adults, approximately 500 individuals ages 18-64 and 250 individuals greater than or equal to age 65. Study procedures include: physical exam, blood samples, completing a memory aid to record vaccine side effects, medications and daily oral temperature. Participants will be involved in study related procedures for up to 13 months.

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread prompting the World Health Organization to declare a pandemic. Data from several cohorts in different age groups that received licensed trivalent seasonal influenza vaccines suggest that these vaccines are unlikely to provide protection against the new virus. These data indicate the need to develop vaccines against the new H1N1 strain and suggest that different vaccine strategies (e.g., number of doses, need for adjuvant) may be appropriate for persons in different age groups. Based on clinical data from the clinical trials with vaccines containing novel influenza A antigens, a higher dosage, or multiple doses of a novel antigen may be necessary to generate potentially protective antibody responses. Alternatively, inactivated influenza H1N1 vaccines administered with adjuvants, such as AS03, may confer protection to a maximal number of vaccine recipients. This protocol will explore antibody responses following vaccination with an inactivated influenza H1N1 virus vaccine at 3 different dose levels combined with AS03 adjuvant and at 2 different dose levels administered without adjuvant. This study will assess the immune response following a single dose of vaccine with or without AS03 adjuvant, to assess whether individuals have any pre-existing 'prime' immunity, such that the initial H1N1 vaccination serves as a boost, thus conferring a more rapid time to protection with the need for fewer doses. Antibody responses will be assessed 8 days after each dose to evaluate the development of an anamnestic response. In addition, antibody responses will be assessed 21 days after each dose. The primary objectives are: safety, to assess the safety of inactivated H1N1 vaccine when administered at 3.75, 7.5 or 15 mcg combined with AS03 adjuvant and at 7.5 or 15 mcg administered without adjuvant; and immunogenicity, to assess the antibody response at Day 21 following a single dose of inactivated H1N1 vaccine when administered at 3.75, 7.5 or 15 mcg combined with AS03 adjuvant and at 7.5 or 15 mcg administered without adjuvant, stratified by age of recipient. The secondary objective is immunogenicity, to assess the antibody response following 2 doses of inactivated H1N1 vaccine when administered at 3.75, 7.5 or 15 mcg combined with AS03 adjuvant and at 7.5 or 15 mcg administered without adjuvant, stratified by age of recipient. Participants will include up to 800 healthy adults who have no history of novel influenza H1N1 2009 infection or novel influenza H1N1 2009 vaccination. This is a randomized, double-blinded, Phase II study. Subjects will be randomized into 5 groups, stratified by age (150 subjects per dose group with 100 subjects in the 18-64 years of age stratum and 50 subjects in the greater than or equal to 65 years of age stratum), to receive intramuscular inactivated influenza H1N1 vaccine at 3.75, 7.5 or 15 mcg combined with AS03 adjuvant (Groups 1, 2, and 3, respectively) or at 7.5 or 15 mcg without adjuvant (Groups 4 and 5, respectively). The vaccine, with and without adjuvant, will be administered at Days 0 and 21. Following immunization, safety will be measured by assessment of adverse events (AEs) through 21 days following the last vaccination (Day 42 for those receiving both doses and Day 21 for those who do not receive the second dose), serious adverse events (SAEs) and new-onset chronic medical conditions through 12 months post final vaccination (Day 365 after second vaccination), and reactogenicity to the vaccine for 8 days following each vaccination (Day 0-7). Immunogenicity testing will include hemagglutination inhibition assay (HAI) and neutralizing antibody testing on serum obtained prior to each vaccination, 8-10 days after each vaccination, 21 days (Day 42), 6 months (Day 201) and 12 months (Day 386) following the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Are males or non-pregnant females age 18 and older, inclusive.
* Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for greater than or equal to 1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods during the study for at least 30 days following the last vaccination.
* Are in good health, as determined by vital signs, medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and limited physical examination. A stable chronic medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company etc, or that is done for financial reasons, as long as in the same class of medication will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome will not be considered a violation of this inclusion criterion.
* Have erythrocyte sedimentation rate (ESR) less than 30 mm per hour.
* Are able to understand and comply with planned study procedures.
* Provide written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Have a known allergy to eggs or other components of the vaccine (including squalene based adjuvants, thimerosal, neomycin, polymyxin, and chicken protein).
* Have a positive urine or serum pregnancy test within 24 hours prior to vaccination if female of childbearing potential or women who are breastfeeding.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have long term use of glucocorticoids including oral, parenteral or high-dose inhaled steroids (>800 micrograms (mcg)/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed.)
* Have a diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis.
* Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
* Are receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study (prior to the Day 386 clinic visit - 365 days after the second vaccination).
* Have received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following the second vaccination. This is inclusive of seasonal influenza vaccines.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, or would interfere with the evaluation of responses.
* Have a history of severe reactions following previous immunization with influenza virus vaccines.
* Have an acute illness, including an oral temperature greater than 100.4 degrees Fahrenheit, within 3 days prior to vaccination.
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Participated in a novel influenza H1N1 2009 vaccine study in the past 2 years or have a history of novel influenza H1N1 2009 infection prior to enrollment.
* Have known active human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C infection or autoimmune hepatitis.
* Have a history of alcohol or drug abuse in the last 5 years.
* Plan to travel outside of North America in the time between the first vaccination and 42 days following the first vaccination.
* Have a history of Guillain-Barré Syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Safety: occurrence of safety laboratory adverse events (AEs). | Days 0, 8-10, 21 and 29.
Safety: occurrence of vaccine-associated serious adverse events (SAEs). | Throughout the course of the study.
Immunogenicity: proportion of subjects, stratified by age, achieving a serum HAI antibody titer of 1:40 or greater, against influenza H1N1 2009 virus at Day 21 following a single dose of H1N1 vaccine combined with or without AS03 adjuvant. | Day 21.
Immunogenicity: proportion of subjects, stratified by age, with 4-fold or greater hemagglutination inhibition (HAI) antibody titer increases against influenza H1N1 2009 virus at Day 21 following a single dose of H1N1 vaccine with or without AS03. | Day 21.
Safety: occurrence of solicited local and systemic adverse events (AEs). | Within 8 days post vaccination (Day 0-7).

SECONDARY OUTCOMES:
Immunogenicity: proportion of subjects, stratified by age, achieving a serum HAI antibody titer of 1:40 or greater against influenza H1N1 2009 virus following 2 doses of H1N1 vaccine combined with or without AS03 adjuvant. | Day 29, Day 42, 6 months (Day 201) and 12 months (Day 386).
Immunogenicity: proportion of subjects, stratified by age, with 4-fold or greater HAI antibody titer increases against influenza H1N1 2009 virus following 2 doses of H1N1 vaccine combined with or without AS03 adjuvant. | Day 29, Day 42, 6 months (Day 201) and 12 months (Day 386).